CLINICAL TRIAL: NCT05539612
Title: Binah.ai Visual Vitals Application - Validation Study
Status: Completed | Type: Observational
Sponsor: Binah.ai LTD. (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-455
Record Dates: First submitted 2022-09-11; First posted 2022-09-14 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Respiratory and Pulse Rate Accuracy Validation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to conduct a Respiratory and Pulse Rate accuracy validation comparing the Binah.ai Visual Vitals Application to the Reference, an FDA cleared End Tidal Carbon Dioxide monitor (GE Datex-Ohmeda), and a standard ECG reference (respectively).

ELIGIBILITY:
Inclusion Criteria:

* Subject must have the ability to understand and provide written informed consent
* Subject must be ≥18 years of age
* Subject must be willing and able to comply with study procedures and duration

Exclusion Criteria:

* Subjects who refuse or are unable to provide to sign an informed written consent for study
* Participants evaluated by the Investigator and Clinical Staff and found to be medically unsuitable or have self-reported health conditions that are currently unstable as identified in the Health Assessment Form and Health Screening
* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor Region Of Interest (ROI) which would limit the ability to test ROI needed for the study.

Tattoo in the optical path which would limit the ability to test ROI needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular areas utilized.)

* Subjects with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, or other medical sensors (self-reported)
* Other known health condition, should be considered upon disclosure in health assessment form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is carefully designed to represent the intended population for the intended use of the Binah.ai Visual Vitals Application. The study population will be comprised of diversity in race, age, gender, BMI, skin tone, and health conditions. The health conditions will constitute certain proportions of healthy controls (to allow testing over the full range of breaths per minute) and disease comorbidities (to represent comorbidities such as COPD, CHF, Asthma, Diabetes, Hypertension, Diabetes and Obesity).
  The goal is to include a range of skin pigmentations, including at least 5 darkly pigmented subjects or 15% of the subject pool, whichever is larger.
  Subject enrollment and participation in this clinical study is based on meeting the inclusion criteria and none of the exclusion criteria, a satisfactory health screen, and the subject and data demographics needed for the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Respiratory Rate accuracy validation | From admission to discharge, up to 2 hours
  Respiratory Rate accuracy validation comparing the Binah.ai Visual Vitals Application to the Reference, an FDA cleared End Tidal Carbon Dioxide monitor (GE Datex-Ohmeda).
Pulse Rate accuracy validation | From admission to discharge, up to 2 hours
  Pulse Rate accuracy validation comparing the Binah.ai Visual Vitals Application to the Reference, a standard ECG.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinimark, LLC, Louisville, Colorado, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/12/NCT05539612/ICF_000.pdf